CLINICAL TRIAL: NCT01946594
Title: Pilot Study to Assess the Effect of Prophylactic Antipyretics on Immune Responses and Rates of Fever After 2013-2014 Inactivated Influenza Vaccine (IIV) in Young Children
Brief Title: Clinical Immunization Safety Assessment (CISA) Project: Pilot Study to Assess the Effect of Prophylactic Antipyretics on Immune Responses and Fever After IIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00048541; 200-2012-53663 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2013-09-17; First posted 2013-09-19 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Fever
Keywords: fever; antipyretics; acetaminophen; influenza vaccine; influenza, human; body temperature changes; Orthomyxoviridae Infections; RNA virus infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases
MeSH Terms: conditions — Fever; Influenza, Human; Body Temperature Changes; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen Arm (Active Comparator): Acetaminophen Suspension 160 mg / 5 mL:
  Oral dose immediately following IIV and every 4-6 hours up to 24 hours (Maximum 5 oral doses)
  Interventions: Other: Acetaminophen
- Placebo Arm (Placebo Comparator): Placebo Suspension:
  Oral dose immediately following IIV and every 4-6 hours up to 24 hours (Maximum 5 oral doses)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Acetaminophen
  Arms: Acetaminophen Arm
Other: Placebo
  Arms: Placebo Arm

SUMMARY:
The study team aims to conduct a double-blind, placebo-controlled, pilot study to assess the effect of prophylactic antipyretics on the immune responses and rates of fever after inactivated influenza vaccine (IIV) in children 12 through 35 months of age. In this pilot, 40 healthy children, 12 through 35 months of age, including some children at risk of febrile seizure, will be randomized to receive prophylactic acetaminophen or oral placebo immediately following and every 4 to 6 hours in the 24 hours after receipt of a dose of IIV. Data derived from the pilot study will be used to assess the feasibility of conducting a larger scale study. Feasibility will include assessments of the speed and ease of study recruitment and adherence to and completion of study assessments. Children will be followed for the occurrence of fever, fussiness, changes in appetite and sleep patterns, and use of medical services on the day of and day following vaccination. Antibody to influenza antigens contained in the 2013-2014 vaccine as measured by hemagglutination inhibition (HAI) antibody will be assessed at baseline and four weeks following vaccination. The proportions of children experiencing fever, having solicited reactions, using medical services, demonstrating a serologic response corresponding to seroprotection and seroconversion to each of the IIV antigens will be determined for groups of children receiving acetaminophen and placebo. Likewise geometric mean HAI titers (GMT) and corresponding 95% confidence intervals for each IIV antigen will be calculated for both vaccine groups.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in the study the following enrollment criteria must be met:

1. The child must be 12 through 35 months of age.
2. The child must only need a single dose of IIV during the current season. (Children only need 1 dose of vaccine in 2013-14 if they received a total of 2 or more doses of seasonal vaccine since July 1, 2010. Children who did not receive a total of 2 or more doses of seasonal vaccine since July 1, 2010 require 2 doses in 2013-14).[19]
3. The parent/guardian must be willing and capable of providing written informed consent for the child.
4. The parent/guardian must be available for follow-up and must at minimum have telephone access.
5. The parent/guardian must agree to sign a medical release for the child so that study personnel may obtain medical information about the child's health (if needed).

Exclusion Criteria:

Participants must not have any of the following:

1. History of receipt of current year's licensed influenza vaccine.
2. History of a severe allergic reaction (e.g. anaphylaxis) to any component of influenza vaccine, including egg protein, formaldehyde, octylphenol ethoxylate, gelatin, or thimerosal if using thimerosal containing vaccine.
3. History of a severe allergic reaction (e.g. anaphylaxis) following a prior dose of influenza vaccine.
4. History of an allergic reaction following acetaminophen or ingredients in the acetaminophen product.
5. History of an allergic reaction following ibuprofen or ingredients in the ibuprofen product.
6. History of liver disease.
7. Currently taking the blood thinning drug warfarin (Coumadin).
8. Received any other licensed vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to vaccination in this study or expects to receive a licensed vaccine during the 28 days following the last vaccination in this study. Concomitant vaccinations are not allowed.
9. Routine immunizations are delayed or will be delayed by not being able to receive a concomitantly administered vaccine or a needed vaccine in the 28 days following receipt of the influenza vaccine.
10. Received an experimental/investigational agent (vaccine, drug, biologic, device, blood product, or medication) within 28 days prior to vaccination in this study, or expects to receive an experimental/investigational agent within the follow-up time period (28 days after the last vaccination in this study).
11. A moderate to severe acute illness and/or a reported temperature greater than or equal to 100.0°F (37.8°C) within 72 hours prior to first dose of IIV or an axillary temperature greater than or equal to 100.0°F (37.8°C) at the time of enrollment. (This may result in a temporary delay of vaccination).
12. Receipt of an antipyretic medication (acetaminophen or ibuprofen) within 72 hours prior to the first dose of IIV (This may result in a temporary delay of vaccination) or is already planning to administer a prophylactic antipyretic medication on the day of and the day following IIV (this exclusion does not apply if the caretaker indicates he/she might administer antipyretics after vaccination to reduce a fever).
13. Immunosuppression as a result of an underlying illness or treatment, or use of anti-cancer chemotherapy or radiation therapy within the preceding 36 months.
14. Long term (at least 14 days of prednisone 2 mg/kg/day or equivalent other glucocorticoid), any parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (topical and nasal steroids are allowed).
15. History of Guillain-Barré syndrome within 6 weeks of a prior dose of influenza vaccine.
16. Has any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Completion of study procedures | 1 month
  Percent of participants for whom study procedures were completed successfully (prophylactic medication administered, temperature measured, memory aid completed, venipunctures performed)

SECONDARY OUTCOMES:
Immune Response to IIV | 1 month
  Immune responses (hemagglutination inhibition assay) to IIV in each group (proportion of subjects demonstrating seroprotection and seroconversion and geometric mean titer)

OTHER OUTCOMES:
IIV reactogenicity and use of medical care services | 2 days
  Proportion of subjects in each group with fever, fussiness, change in appetite or sleep patterns, and receipt of medical attention

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel B Walter, MD, Principal Investigator — Duke University; Karen Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Duke University Health System, Durham, North Carolina, United States